CLINICAL TRIAL: NCT04071795
Title: Clinical Reminder Changes to Increase Smoking Cessation Treatment in Outpatient Psychiatry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00813
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: 2 arm cluster randomized study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opt Out (Experimental): Training and Academic Detailing
  Interventions: Behavioral: Opt-Out Reminder
- Opt In (Experimental): Training and Academic Detailing
  Interventions: Behavioral: Opt-In Reminder

INTERVENTIONS:
Behavioral: Opt-Out Reminder — half will receive a clinical reminder that includes a standing NRT order and a referral to cessation counseling that will automatically generate unless the provider actively opts-out
  Arms: Opt Out
Behavioral: Opt-In Reminder — Half of the psychiatrists will receive a reminder that encourages the psychiatrist to offer cessation medications and referral to cessation counseling to patients interested in quitting
  Arms: Opt In

SUMMARY:
This study will use a scientifically robust, mixed-methods, two-arm cluster-randomized study design. Investigators will implement a tobacco use clinical reminder for outpatient psychiatrists practicing at the VA New York Harbor Healthcare System (N = 20). Half of the psychiatrists will receive a reminder that encourages the psychiatrist to offer cessation medications and referral to cessation counseling to patients interested in quitting (Opt-In Reminder). The other half will receive a clinical reminder that includes a standing nicotine replacement therapy (NRT) order and a referral to cessation counseling that will automatically generate unless the provider actively opts-out (Opt-Out Reminder). Prior to implementation of the reminders, psychiatrists in both arms will receive a one-hour training on tobacco treatment and individual education outreach to demonstrate the clinical reminder and answer questions (academic detailing).

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrists
* Works in outpatient psychiatry at Manhattan or Brooklyn VA campus and has no plans to leave in the next 6 months
* Patient Post-Visit Survey Population
* Had a visit with a psychiatrist included in the study Current smoker

Exclusion Criteria:

* Outpatient Psychiatrists:
* None
* Patient Post-Visit Survey Population:
* Non-English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rogers, DrPH, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Derived] Rogers ES, Wysota C, Prochaska JJ, Tenner C, Dognin J, Wang B, Sherman SE. A behavioral economic intervention to increase psychiatrist adherence to tobacco treatment guidelines: a provider-randomized study protocol. Implement Sci Commun. 2020;1:32. doi: 10.1186/s43058-020-00011-x. Epub 2020 Feb 25. PMID 32617528

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, psychiatrists practicing at the VA New York Harbor Healthcare System were enrolled and randomized to either the Opt-Out Reminder group (n=58) or Opt-In Reminder group (n=82).
  A waiver of informed consent was granted to extract data on patients (Opt-Out Reminder, n=240; Opt-In Reminder, n=303) who were seen by the participating psychiatrists. These patients were not considered to be enrolled participants
Groups:
- Opt Out Reminder - Psychiatrists: Psychiatrists in the Opt-Out Reminder group received a clinical reminder that included a standing nicotine replacement therapy (NRT) order and a referral to cessation counseling that automatically generated unless the provider actively opted-out.
- Opt-Out Reminder - Patients: Patients of psychiatrists randomized to the opt-out reminder arm.
- Opt In Reminder - Psychiatrists: Psychiatrists in the Opt-In Reminder group received a reminder that encouraged the psychiatrist to offer cessation medications and referral to cessation counseling to patients interested in quitting.
- Opt In Reminder - Patients: Patients of psychiatrists randomized to the opt-in reminder arm.
Period: Overall Study
Arm/Group | Opt Out Reminder - Psychiatrists | Opt-Out Reminder - Patients | Opt In Reminder - Psychiatrists | Opt In Reminder - Patients
Started | 58 | 240 | 82 | 303
Completed | 34 | 240 | 55 | 303
Not Completed | 24 | 0 | 27 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were only collected from participating psychiatrists. A waiver of informed consent was granted to extract data on patients who were seen by the participating psychiatrists. No baseline data were collected for these patients.
Groups:
- Opt Out Reminder: Psychiatrists in the Opt-Out Reminder group received a clinical reminder that included a standing nicotine replacement therapy (NRT) order and a referral to cessation counseling that automatically generated unless the provider actively opted-out.
- Opt In Reminder: Psychiatrists in the Opt-In Reminder group received a reminder that encouraged the psychiatrist to offer cessation medications and referral to cessation counseling to patients interested in quitting.
- Total: Total of all reporting groups
Arm/Group | Opt Out Reminder | Opt In Reminder | Total
Number analyzed (Participants) | 34 | 55 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (16.8) | 66.6 (9.23) | 64.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 32 | 49 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 23 | 45 | 68
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 16 | 23 | 39
  White | 9 | 19 | 28
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 34 | 55 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Screened for Smoking
Description: Number of patients with documented current smoking in the medical record who were screened for tobacco use during their psychiatry visit. Data derived from medial records.
Time Frame: Up to Month 6
Population: A waiver of HIPAA authorization was granted to abstract patient electronic health record (EHR) data from VA administrative data for the purposes of analysis of the primary outcomes. The overall number of participants analyzed represents patients (Participants) with available EHR data (Opt-Out Reminder Group, n = 240; Opt-In Reminder Group = 303) who visited a participating psychiatrist.
Measure: Count of Participants; unit: Participants
Groups:
- Opt-Out Reminder - Patients of Participating Psychiatrists: Mental health patients with documented current smoking in the medical record who visited a psychiatrist randomized to receive the Opt-Out reminder.
- Opt-In Reminder - Patients of Participating Psychiatrists: Mental health patients with documented current smoking in the medical record who visited a psychiatrist randomized to receive the Opt-In reminder.
Arm/Group | Opt-Out Reminder - Patients of Participating Psychiatrists | Opt-In Reminder - Patients of Participating Psychiatrists
Number analyzed (Participants) | 240 | 303
Participants | 240 | 303

2. Primary Outcome: Number of Smokers Prescribed a Cessation Medication
Description: Number of people with documented current smoking in the medical record who were prescribed cessation medication.
Time Frame: Up to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Opt-Out Reminder - Patients of Participating Psychiatrists | Opt-In Reminder - Patients of Participating Psychiatrists
Number analyzed (Participants) | 240 | 303
Participants | 63 | 47

3. Primary Outcome: Number of Smokers Referred to Counseling
Description: Number of people with documented current smoking in the medical record for whom counseling referrals were ordered.
Time Frame: Up to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Opt-Out Reminder - Patients of Participating Psychiatrists | Opt-In Reminder - Patients of Participating Psychiatrists
Number analyzed (Participants) | 240 | 303
Participants | 59 | 24

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Adverse Event/Serious Adverse Events/All-Cause Mortality data were collected only for participating psychiatrists. AE/SAE/All-Cause Mortality data were not collected for Participants with extracted outcome measure data who visited the participating psychiatrists. Thus, the number of participants analyzed for AEs/SAEs/All-Cause Mortality in the Opt-Out Reminder and Opt-In Reminder arms is 34 and 55, respectively (equal to the number of psychiatrists who completed the trial in each arm).
Arm/Group | Opt Out Reminder | Opt In Reminder
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/55
Other Adverse Events (participants affected / at risk) | 0/34 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04071795/Prot_SAP_000.pdf